CLINICAL TRIAL: NCT06326996
Title: Thiamine Intervention and Cognition in Older Adults Undergoing Coronary Artery Bypass Grafting - A Randomized Clinical Trial.
Brief Title: Thiamine Intervention and Coronary Artery Bypass Grafting
Acronym: B1&CABG
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rajesh Kumar, PhD, Professor of Anesthesiology and Radiological Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-001185; R21AG081720-01A1 (NIH)
Record Dates: First submitted 2024-03-07; First posted 2024-03-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Coronary Heart Disease; Coronary Artery Bypass Grafting
Keywords: thiamine intervention
MeSH Terms: conditions — Coronary Disease | interventions — Thiamine

STUDY DESIGN:
Intervention Model Description: Post-CABG patients with and without thiamine treatment.
Who Masked: Participant
Masking Description: Participants will be assigned a random number, double-blind randomized, & longitudinal study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Post-CABG patients with Thiamine Treatment Intervention. (Experimental): Assess cognition and evaluate blood thiamine, lactate, and inflammatory marker levels in patients receiving thiamine intervention treatment within 5 days (baseline) and one month after CABG.
  Interventions: Drug: Thiamine
- Post-CABG patients without Thiamine Treatment Intervention. (Placebo Comparator): Assess cognition and evaluate blood thiamine, lactate, and inflammatory marker levels in patients receiving placebo treatment within 5 days (baseline) and one month after CABG.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thiamine — Participants will be given an infusion of thiamine.
  Other Names: Vitamin B1
  Arms: Post-CABG patients with Thiamine Treatment Intervention.
Drug: Placebo — Participants will be given an infusion of the placebo treatment.
  Other Names: inactive
  Arms: Post-CABG patients without Thiamine Treatment Intervention.

SUMMARY:
The purpose of this study is to gain a better understanding of the association between brain changes and cognitive deficits in coronary heart disease (CHD) patients undergoing coronary artery bypass grafting (CABG) and whether a low-cost thiamine intervention can be used to reduce post-CABG cognitive issues in CHD subjects.

DETAILED DESCRIPTION:
Using a two-group, double-blind randomized, longitudinal study design, 52 coronary heart disease (CHD) patients undergoing coronary artery bypass grafting (CABG) (ages 60-80 years; 26 thiamine treatment and 26 placebo) will participate in cognitive assessment and evaluation of blood thiamine, lactate, and inflammatory marker levels. The investigators propose that thiamine infusion will help in reducing lactate and inflammatory marker levels, as observed in other conditions. The findings from this study might serve as a novel and innovative treatment strategy for protection against declining cognition, and hence better outcomes, and improved quality of life and daily activities. This clinical trial study will provide required data regarding the benefits of a low-cost thiamine intervention that could be implemented on a large-scale clinical trial to reduce post-CABG cognitive deficits in older CHD, and thus, decrease early dementia, improve social function, increase quality of life and daily activities, and reduce healthcare costs in this serious older CHD patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Coronary Heart Disease (CHD) scheduled for Bypass Grafting (CABG)
* Thiamine deficiency before CABG
* European System for Cardiac Operative Risk Evaluation II (EuroSCORE II) >1.5%
* Off-pump surgery

Exclusion Criteria:

* Dementia at baseline [Montreal Cognitive Assessment (MoCA) <21 within 5 days before CABG]
* Current in-take of thiamine
* Known thiamine allergy
* Uncontrolled blood glucose levels
* Unable to give consent due to illness
* History of hyperlactatemia
* Recent (within several years and/or up to the judgment of the PI/co-PIs) cerebral incidents (seizure or head trauma resulting in loss of consciousness and/or concussion)
* Stroke
* Diagnosed psychiatric diseases (clinical depression, schizophrenia, manic-depression)
* Patients with history of alcohol or substance abuse
* Acute or chronic infections (tuberculosis, hepatitis, or encephalopathy)
* Diagnosed neuro-degenerative diseases (Alzheimer's or Parkinson's disease)
* Chronic immunodeficiency (including HIV)
* Congenital brain deficits will also be excluded

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Effects of thiamine treatment intervention on blood lactate levels. | Baseline and after 1 month after CABG.
  Assess thiamine treatment effect on blood lactate levels in CABG patients with and without intervention measured via blood gas analyzer (ABL90 flex plus, Radiometer).
Effects of thiamine treatment intervention on blood thiamine levels. | Baseline and after 1 month after CABG.
  Assess thiamine treatment effect on blood thiamine levels in CABG patients with and without intervention measured via blood gas analyzer (ABL90 flex plus, Radiometer).
Effects of thiamine treatment intervention on blood inflammatory levels. | Baseline and after 1 month after CABG.
  Assess thiamine treatment effect on blood inflammatory levels in CABG patients with and without intervention measured via a custom kit, including cytokines from the human 38-plex magnetic cytokine/chemokine kit, will be used per manufacturer's instructions.
Evaluate cognitive function in CABG patients with thiamine treatment. | Baseline and after 1 month after CABG.
  The investigators will evaluate cognitive function using the NIH Toolbox Cognition Battery (executive function, attention, and speed). CABG patients with thiamine treatment will show a change in cognition over CABG patients without thiamine treatment.
Evaluate long term effects of thiamine treatment intervention on cognitive function in CABG patients with thiamine treatment. | 6 months after CABG.
  The investigators will evaluate cognitive function using the NIH Toolbox Cognition Battery (executive function, attention, and speed). CABG patients with thiamine treatment will show a change in cognition over CABG patients without thiamine treatment.
Examine cognition in CABG patients with thiamine treatment. | Baseline and 1 month after CABG.
  The investigators will examine cognition using the Wide Range Assessment of Memory and Learning 2 (WRAML2). CABG patients with thiamine treatment will show a change in cognition over CABG patients without thiamine treatment.
Examine long term effects of thiamine treatment intervention on cognition in CABG patients with thiamine treatment. | 6 months after CABG.
  The investigators will examine cognition using the Wide Range Assessment of Memory and Learning 2 (WRAML2). CABG patients with thiamine treatment will show a change in cognition over CABG patients without thiamine treatment.
Cognition assessment in CABG patients after thiamine treatment. | Baseline and 1 month after CABG.
  The investigators will assess cognition using the Montreal Cognitive Assessment (MoCA). CABG patients with thiamine treatment will show a change in cognition over CABG patients without thiamine treatment. The MoCA is a brief cognitive assessment administered to the participant by the investigator. The score ranges from 0 to 30, with higher scores indicating better cognitive function.
Assessment of long term effects of thiamine treatment intervention on cognition in CABG patients after thiamine treatment. | 6 months after CABG.
  The investigators will assess cognition using the Montreal Cognitive Assessment (MoCA). CABG patients with thiamine treatment will show a change in cognition over CABG patients without thiamine treatment. The MoCA is a brief cognitive assessment administered to the participant by the investigator. The score ranges from 0 to 30, with higher scores indicating better cognitive function.
Long term effect of thiamine treatment intervention on quality of life. | 6 months after CABG.
  Examine the long-term quality of life in older CHD subjects with and without thiamine intervention treatment as measured by NIH validated Short-Form 36 (SF-36) survey. The SF-36 is a 36 question form filled out by the participant and scored by the investigator. The score ranges from 0 to 100, with higher scores indicating better health status.
Long term effect of thiamine treatment intervention on daily activities using PASE. | 6 months after CABG.
  Examine the long-term daily activities status in older CHD subjects with and without thiamine intervention treatment as measured by NIH validated Physical Activity Scale for the Elderly (PASE). PASE is a brief self-administered questionnaire measuring physical activity which generates a score, ranging from 0 to 793, with higher scores indicating greater physical activity.
Long term effect of thiamine treatment intervention on daily activities using PPA. | 6 months after CABG.
  Examine the long-term daily activities status in older CHD subjects with and without thiamine intervention treatment as measured by Paffenbarger Physical Activity (PPA).

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Kumar, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make every effort to publish data in a timely manner. Once the findings related to changes in blood lactate, thiamine, and inflammatory levels based on blood pathology and cognition assessment data before and after thiamine intervention on CHD subjects before and after CABG have been published or by the end of award performance period, whichever is sooner, the blood levels, cognitive data, demographics, mood, and clinical data (devoid of individual identifiers) will be deposited in NIH supported domain-specific data sharing repository (NIMH Data Archive). All data will be labeled with consistent unique identifiers that will make it easily findable in data repository to interested research investigators. Data will be available forever after sharing with data repository to other investigators for secondary analyses.
Time Frame: Once the findings have been published or by the end of award performance period, whichever is sooner.
Access Criteria: Any research investigator

REFERENCES:
- [Background] Gershon RC, Wagster MV, Hendrie HC, Fox NA, Cook KF, Nowinski CJ. NIH toolbox for assessment of neurological and behavioral function. Neurology. 2013 Mar 12;80(11 Suppl 3):S2-6. doi: 10.1212/WNL.0b013e3182872e5f. PMID 23479538
- [Background] Hodes RJ, Insel TR, Landis SC; NIH Blueprint for Neuroscience Research. The NIH toolbox: setting a standard for biomedical research. Neurology. 2013 Mar 12;80(11 Suppl 3):S1. doi: 10.1212/WNL.0b013e3182872e90. PMID 23479536
- [Background] Sheslow DA, W. . Wide range assessment of memory and learning (2nd edition) administration and technical manual In: Editor, ed.^eds. Wide range assessment of memory and learning (2nd edition) administration and technical manual. City: Psychological Assessment Resources, 2003.
- [Background] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Bauer PJ, Carlozzi NE, Slotkin J, Blitz D, Wallner-Allen K, Fox NA, Beaumont JL, Mungas D, Nowinski CJ, Richler J, Deocampo JA, Anderson JE, Manly JJ, Borosh B, Havlik R, Conway K, Edwards E, Freund L, King JW, Moy C, Witt E, Gershon RC. Cognition assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S54-64. doi: 10.1212/WNL.0b013e3182872ded. PMID 23479546
- [Background] Ware J, Kosinski M, Dewey JE. How to score version 2 of the SF- 36 health survey. Lincoln, RI: QualityMetric Incorporated; 2000 p 229: 2000.
- [Background] Washburn RA, Smith KW, Jette AM, Janney CA. The Physical Activity Scale for the Elderly (PASE): development and evaluation. J Clin Epidemiol. 1993 Feb;46(2):153-62. doi: 10.1016/0895-4356(93)90053-4. PMID 8437031
- [Background] Bolszak S, Casartelli NC, Impellizzeri FM, Maffiuletti NA. Validity and reproducibility of the Physical Activity Scale for the Elderly (PASE) questionnaire for the measurement of the physical activity level in patients after total knee arthroplasty. BMC Musculoskelet Disord. 2014 Feb 20;15:46. doi: 10.1186/1471-2474-15-46. PMID 24555852
- [Background] Paffenbarger RS Jr, Wing AL, Hyde RT. Physical activity as an index of heart attack risk in college alumni. Am J Epidemiol. 1978 Sep;108(3):161-75. doi: 10.1093/oxfordjournals.aje.a112608. PMID 707484
- [Background] Hall MJ, DeFrances CJ, Williams SN, Golosinskiy A, Schwartzman A. National Hospital Discharge Survey: 2007 summary. Natl Health Stat Report. 2010 Oct 26;(29):1-20, 24. PMID 21086860
- [Background] Frost L, Molgaard H, Christiansen EH, Hjortholm K, Paulsen PK, Thomsen PE. Atrial fibrillation and flutter after coronary artery bypass surgery: epidemiology, risk factors and preventive trials. Int J Cardiol. 1992 Sep;36(3):253-61. doi: 10.1016/0167-5273(92)90293-c. PMID 1358829
- [Background] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Background] Silber JH, Rosenbaum PR, Schwartz JS, Ross RN, Williams SV. Evaluation of the complication rate as a measure of quality of care in coronary artery bypass graft surgery. JAMA. 1995 Jul 26;274(4):317-23. PMID 7609261
- [Background] Newman MF, Kirchner JL, Phillips-Bute B, Gaver V, Grocott H, Jones RH, Mark DB, Reves JG, Blumenthal JA; Neurological Outcome Research Group and the Cardiothoracic Anesthesiology Research Endeavors Investigators. Longitudinal assessment of neurocognitive function after coronary-artery bypass surgery. N Engl J Med. 2001 Feb 8;344(6):395-402. doi: 10.1056/NEJM200102083440601. PMID 11172175
- [Background] Selnes OA, Goldsborough MA, Borowicz LM, McKhann GM. Neurobehavioural sequelae of cardiopulmonary bypass. Lancet. 1999 May 8;353(9164):1601-6. doi: 10.1016/S0140-6736(98)07576-X. PMID 10334272
- [Background] Evered LA, Silbert BS, Scott DA, Maruff P, Ames D. Prevalence of Dementia 7.5 Years after Coronary Artery Bypass Graft Surgery. Anesthesiology. 2016 Jul;125(1):62-71. doi: 10.1097/ALN.0000000000001143. PMID 27127919
- [Background] Kuzma E, Airdrie J, Littlejohns TJ, Lourida I, Thompson-Coon J, Lang IA, Scrobotovici M, Thacker EL, Fitzpatrick A, Kuller LH, Lopez OL, Longstreth WT Jr, Ukoumunne OC, Llewellyn DJ. Coronary Artery Bypass Graft Surgery and Dementia Risk in the Cardiovascular Health Study. Alzheimer Dis Assoc Disord. 2017 Apr-Jun;31(2):120-127. doi: 10.1097/WAD.0000000000000191. PMID 28263191
- [Background] Bjorklund E, Nielsen SJ, Hansson EC, Karlsson M, Wallinder A, Martinsson A, Tygesen H, Romlin BS, Malm CJ, Pivodic A, Jeppsson A. Secondary prevention medications after coronary artery bypass grafting and long-term survival: a population-based longitudinal study from the SWEDEHEART registry. Eur Heart J. 2020 May 1;41(17):1653-1661. doi: 10.1093/eurheartj/ehz714. PMID 31638654
- [Background] Lee TA, Wolozin B, Weiss KB, Bednar MM. Assessment of the emergence of Alzheimer's disease following coronary artery bypass graft surgery or percutaneous transluminal coronary angioplasty. J Alzheimers Dis. 2005 Aug;7(4):319-24. doi: 10.3233/jad-2005-7408. PMID 16131734
- [Background] Thornton EW, Groom C, Fabri BM, Fox MA, Hallas C, Jackson M. Quality of life outcomes after coronary artery bypass graft surgery: relationship to neuropsychologic deficit. J Thorac Cardiovasc Surg. 2005 Oct;130(4):1022-7. doi: 10.1016/j.jtcvs.2005.05.020. PMID 16214514
- [Background] Jabbari A, Banihashem N, Alijanpour E, Vafaey HR, Alereza H, Rabiee SM. Serum lactate as a prognostic factor in coronary artery bypass graft operation by on pump method. Caspian J Intern Med. 2013 Spring;4(2):662-6. PMID 24009956
- [Background] Andersen LW, Liu X, Peng TJ, Giberson TA, Khabbaz KR, Donnino MW. Pyruvate Dehydrogenase Activity and Quantity Decreases After Coronary Artery Bypass Grafting: a Prospective Observational Study. Shock. 2015 Mar;43(3):250-4. doi: 10.1097/SHK.0000000000000306. PMID 25526377
- [Background] Toraman F, Evrenkaya S, Yuce M, Aksoy N, Karabulut H, Bozkulak Y, Alhan C. Lactic acidosis after cardiac surgery is associated with adverse outcome. Heart Surg Forum. 2004 Apr 1;7(2):E155-9. doi: 10.1532/HSF98.20041002. PMID 15138095
- [Background] Lindsay AJ, Xu M, Sessler DI, Blackstone EH, Bashour CA. Lactate clearance time and concentration linked to morbidity and death in cardiac surgical patients. Ann Thorac Surg. 2013 Feb;95(2):486-92. doi: 10.1016/j.athoracsur.2012.07.020. Epub 2012 Sep 7. PMID 22959571
- [Background] Hajjar LA, Almeida JP, Fukushima JT, Rhodes A, Vincent JL, Osawa EA, Galas FR. High lactate levels are predictors of major complications after cardiac surgery. J Thorac Cardiovasc Surg. 2013 Aug;146(2):455-60. doi: 10.1016/j.jtcvs.2013.02.003. Epub 2013 Mar 15. PMID 23507124
- [Background] Hanstock TL, Mallet PE, Clayton EH. Increased plasma d-lactic acid associated with impaired memory in rats. Physiol Behav. 2010 Dec 2;101(5):653-9. doi: 10.1016/j.physbeh.2010.09.018. Epub 2010 Oct 1. PMID 20888356
- [Background] Pekovich SR, Martin PR, Singleton CK. Thiamine deficiency decreases steady-state transketolase and pyruvate dehydrogenase but not alpha-ketoglutarate dehydrogenase mRNA levels in three human cell types. J Nutr. 1998 Apr;128(4):683-7. doi: 10.1093/jn/128.4.683. PMID 9521628
- [Background] Donnino MW, Cocchi MN, Smithline H, Carney E, Chou PP, Salciccioli J. Coronary artery bypass graft surgery depletes plasma thiamine levels. Nutrition. 2010 Jan;26(1):133-6. doi: 10.1016/j.nut.2009.06.004. PMID 20005469
- [Background] Vacas S, Degos V, Tracey KJ, Maze M. High-mobility group box 1 protein initiates postoperative cognitive decline by engaging bone marrow-derived macrophages. Anesthesiology. 2014 May;120(5):1160-7. doi: 10.1097/ALN.0000000000000045. PMID 24162463
- [Background] Berger M, Terrando N, Smith SK, Browndyke JN, Newman MF, Mathew JP. Neurocognitive Function after Cardiac Surgery: From Phenotypes to Mechanisms. Anesthesiology. 2018 Oct;129(4):829-851. doi: 10.1097/ALN.0000000000002194. PMID 29621031
- [Background] Cruickshank AM, Telfer AB, Shenkin A. Thiamine deficiency in the critically ill. Intensive Care Med. 1988;14(4):384-7. doi: 10.1007/BF00262893. PMID 3136196
- [Background] El-Ansary A, Bhat RS, Al-Daihan S, Al Dbass AM. The neurotoxic effects of ampicillin-associated gut bacterial imbalances compared to those of orally administered propionic acid in the etiology of persistent autistic features in rat pups: effects of various dietary regimens. Gut Pathog. 2015 Mar 22;7:7. doi: 10.1186/s13099-015-0054-4. eCollection 2015. PMID 25852770
- [Background] Morris G, Maes M. Oxidative and Nitrosative Stress and Immune-Inflammatory Pathways in Patients with Myalgic Encephalomyelitis (ME)/Chronic Fatigue Syndrome (CFS). Curr Neuropharmacol. 2014 Mar;12(2):168-85. doi: 10.2174/1570159X11666131120224653. PMID 24669210
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Smith T, Gildeh N, Holmes C. The Montreal Cognitive Assessment: validity and utility in a memory clinic setting. Can J Psychiatry. 2007 May;52(5):329-32. doi: 10.1177/070674370705200508. PMID 17542384
- [Background] Pike NA, Roy B, Gupta R, Singh S, Woo MA, Halnon NJ, Lewis AB, Kumar R. Brain abnormalities in cognition, anxiety, and depression regulatory regions in adolescents with single ventricle heart disease. J Neurosci Res. 2018 Jun;96(6):1104-1118. doi: 10.1002/jnr.24215. Epub 2018 Jan 6. PMID 29315714
- [Background] Cabrera-Mino C, Roy B, Woo MA, Singh S, Moye S, Halnon NJ, Lewis AB, Kumar R, Pike NA. Reduced brain mammillary body volumes and memory deficits in adolescents who have undergone the Fontan procedure. Pediatr Res. 2020 Jan;87(1):169-175. doi: 10.1038/s41390-019-0569-3. Epub 2019 Sep 9. PMID 31499515
- [Background] Noorani S, Roy B, Sahib AK, Cabrera-Mino C, Halnon NJ, Woo MA, Lewis AB, Pike NA, Kumar R. Caudate nuclei volume alterations and cognition and mood dysfunctions in adolescents with single ventricle heart disease. J Neurosci Res. 2020 Oct;98(10):1877-1888. doi: 10.1002/jnr.24667. Epub 2020 Jun 12. PMID 32530059
- [Background] Singh S, Roy B, Pike N, Daniel E, Ehlert L, Lewis AB, Halnon N, Woo MA, Kumar R. Altered brain diffusion tensor imaging indices in adolescents with the Fontan palliation. Neuroradiology. 2019 Jul;61(7):811-824. doi: 10.1007/s00234-019-02208-x. Epub 2019 Apr 30. PMID 31041457
- [Background] Roy B, Woo MA, Wang DJJ, Fonarow GC, Harper RM, Kumar R. Reduced regional cerebral blood flow in patients with heart failure. Eur J Heart Fail. 2017 Oct;19(10):1294-1302. doi: 10.1002/ejhf.874. Epub 2017 May 30. PMID 28560737
- [Background] Park B, Roy B, Woo MA, Palomares JA, Fonarow GC, Harper RM, Kumar R. Lateralized Resting-State Functional Brain Network Organization Changes in Heart Failure. PLoS One. 2016 May 20;11(5):e0155894. doi: 10.1371/journal.pone.0155894. eCollection 2016. PMID 27203600
- [Background] Roy B, Vacas S, Ehlert L, McCloy K, Saggar R, Kumar R. Brain Structural Changes in Patients with Pulmonary Arterial Hypertension. J Neuroimaging. 2021 May;31(3):524-531. doi: 10.1111/jon.12840. Epub 2021 Feb 9. PMID 33565204
- [Background] Fernandes CJ, Martins BC, Jardim CV, Ciconelli RM, Morinaga LK, Breda AP, Hoette S, Souza R. Quality of life as a prognostic marker in pulmonary arterial hypertension. Health Qual Life Outcomes. 2014 Aug 30;12:130. doi: 10.1186/s12955-014-0130-3. PMID 25176512
- [Background] Keogh AM, McNeil KD, Wlodarczyk J, Gabbay E, Williams TJ. Quality of life in pulmonary arterial hypertension: improvement and maintenance with bosentan. J Heart Lung Transplant. 2007 Feb;26(2):181-7. doi: 10.1016/j.healun.2006.11.009. PMID 17258153
- [Background] Muller-Nordhorn J, Roll S, Willich SN. Comparison of the short form (SF)-12 health status instrument with the SF-36 in patients with coronary heart disease. Heart. 2004 May;90(5):523-7. doi: 10.1136/hrt.2003.013995. PMID 15084550
- [Background] Ueno K, Kamiya K, Hamazaki N, Nozaki K, Ichikawa T, Yamashita M, Uchida S, Kawabata M, Maekawa E, Yamaoka-Tojo M, Matsunaga A, Ako J. Usefulness of physical function sub-item of SF-36 survey to predict exercise intolerance in patients with heart failure. Eur J Cardiovasc Nurs. 2022 Mar 3;21(2):174-177. doi: 10.1093/eurjcn/zvab052. PMID 34324626
- [Background] Chatzinikolaou A, Tzikas S, Lavdaniti M. Assessment of Quality of Life in Patients With Cardiovascular Disease Using the SF-36, MacNew, and EQ-5D-5L Questionnaires. Cureus. 2021 Sep 14;13(9):e17982. doi: 10.7759/cureus.17982. eCollection 2021 Sep. PMID 34667665
- [Background] Wallace J, Ceschin R, Lee VK, Beluk NH, Burns C, Beers S, Lo C, Panigrahy A, Badaly D. Psychometric Properties of the NIH Toolbox Cognition and Emotion Batteries Among Children and Adolescents with Congenital Heart Defects. medRxiv [Preprint]. 2023 Feb 14:2023.02.11.23285800. doi: 10.1101/2023.02.11.23285800. PMID 36824875
- [Background] Lee IM, Sesso HD, Paffenbarger RS Jr. Physical activity and coronary heart disease risk in men: does the duration of exercise episodes predict risk? Circulation. 2000 Aug 29;102(9):981-6. doi: 10.1161/01.cir.102.9.981. PMID 10961961
- [Background] Sesso HD, Paffenbarger RS Jr, Lee IM. Physical activity and coronary heart disease in men: The Harvard Alumni Health Study. Circulation. 2000 Aug 29;102(9):975-80. doi: 10.1161/01.cir.102.9.975. PMID 10961960
- [Background] Paffenbarger RS Jr, Hyde RT, Jung DL, Wing AL. Epidemiology of exercise and coronary heart disease. Clin Sports Med. 1984 Apr;3(2):297-318. PMID 6388854
- [Background] Falder S, Silla R, Phillips M, Rea S, Gurfinkel R, Baur E, Bartley A, Wood FM, Fear MW. Thiamine supplementation increases serum thiamine and reduces pyruvate and lactate levels in burn patients. Burns. 2010 Mar;36(2):261-9. doi: 10.1016/j.burns.2009.04.012. Epub 2009 Jun 6. PMID 19501976
- [Background] Lindenbaum GA, Larrieu AJ, Carroll SF, Kapusnick RA. Effect of cocarboxylase in dogs subjected to experimental septic shock. Crit Care Med. 1989 Oct;17(10):1036-40. doi: 10.1097/00003246-198910000-00014. PMID 2791565
- [Background] Bautista-Hernandez VM, Lopez-Ascencio R, Del Toro-Equihua M, Vasquez C. Effect of thiamine pyrophosphate on levels of serum lactate, maximum oxygen consumption and heart rate in athletes performing aerobic activity. J Int Med Res. 2008 Nov-Dec;36(6):1220-6. doi: 10.1177/147323000803600608. PMID 19094430
- [Background] Liu J, Wu JQ, Yang JJ, Wei JY, Gao WN, Guo CJ. Metabolomic study on vitamins B(1), B(2), and PP supplementation to improve serum metabolic profiles in mice under acute hypoxia based on (1)H NMR analysis. Biomed Environ Sci. 2010 Aug;23(4):312-8. doi: 10.1016/S0895-3988(10)60069-4. PMID 20934120
- [Background] Li J, Wynn RM, Machius M, Chuang JL, Karthikeyan S, Tomchick DR, Chuang DT. Cross-talk between thiamin diphosphate binding and phosphorylation loop conformation in human branched-chain alpha-keto acid decarboxylase/dehydrogenase. J Biol Chem. 2004 Jul 30;279(31):32968-78. doi: 10.1074/jbc.M403611200. Epub 2004 May 27. PMID 15166214
- [Background] Barnett SD, Ad N. Surgery for aortic and mitral valve disease in the United States: a trend of change in surgical practice between 1998 and 2005. J Thorac Cardiovasc Surg. 2009 Jun;137(6):1422-9. doi: 10.1016/j.jtcvs.2008.08.071. Epub 2009 Feb 20. PMID 19464459
- [Background] Yusuf S, Zucker D, Peduzzi P, Fisher LD, Takaro T, Kennedy JW, Davis K, Killip T, Passamani E, Norris R, et al. Effect of coronary artery bypass graft surgery on survival: overview of 10-year results from randomised trials by the Coronary Artery Bypass Graft Surgery Trialists Collaboration. Lancet. 1994 Aug 27;344(8922):563-70. doi: 10.1016/s0140-6736(94)91963-1. PMID 7914958
- [Background] Raja PV, Blumenthal JA, Doraiswamy PM. Cognitive deficits following coronary artery bypass grafting: prevalence, prognosis, and therapeutic strategies. CNS Spectr. 2004 Oct;9(10):763-72. doi: 10.1017/s1092852900022409. PMID 15448586
- [Background] Hammon JW Jr, Stump DA, Kon ND, Cordell AR, Hudspeth AS, Oaks TE, Brooker RF, Rogers AT, Hilbawi R, Coker LH, Troost BT. Risk factors and solutions for the development of neurobehavioral changes after coronary artery bypass grafting. Ann Thorac Surg. 1997 Jun;63(6):1613-8. doi: 10.1016/s0003-4975(97)00261-0. PMID 9205158
- [Background] Culley DJ, Flaherty D, Fahey MC, Rudolph JL, Javedan H, Huang CC, Wright J, Bader AM, Hyman BT, Blacker D, Crosby G. Poor Performance on a Preoperative Cognitive Screening Test Predicts Postoperative Complications in Older Orthopedic Surgical Patients. Anesthesiology. 2017 Nov;127(5):765-774. doi: 10.1097/ALN.0000000000001859. PMID 28891828
- [Background] Stroobant N, Van Nooten G, Van Belleghem Y, Vingerhoets G. The effect of CABG on neurocognitive functioning. Acta Cardiol. 2010 Oct;65(5):557-64. doi: 10.1080/ac.65.5.2056243. PMID 21125978
- [Background] Leslie DL, Inouye SK. The importance of delirium: economic and societal costs. J Am Geriatr Soc. 2011 Nov;59 Suppl 2(Suppl 2):S241-3. doi: 10.1111/j.1532-5415.2011.03671.x. PMID 22091567
- [Background] Leslie DL, Marcantonio ER, Zhang Y, Leo-Summers L, Inouye SK. One-year health care costs associated with delirium in the elderly population. Arch Intern Med. 2008 Jan 14;168(1):27-32. doi: 10.1001/archinternmed.2007.4. PMID 18195192
- [Background] Phillips-Bute B, Mathew JP, Blumenthal JA, Grocott HP, Laskowitz DT, Jones RH, Mark DB, Newman MF. Association of neurocognitive function and quality of life 1 year after coronary artery bypass graft (CABG) surgery. Psychosom Med. 2006 May-Jun;68(3):369-75. doi: 10.1097/01.psy.0000221272.77984.e2. PMID 16738066
- [Background] Bursa F, Pleva L. Anaerobic metabolism associated with traumatic hemorrhagic shock monitored by microdialysis of muscle tissue is dependent on the levels of hemoglobin and central venous oxygen saturation: a prospective, observational study. Scand J Trauma Resusc Emerg Med. 2014 Feb 5;22:11. doi: 10.1186/1757-7241-22-11. PMID 24499479
- [Background] Demers P, Elkouri S, Martineau R, Couturier A, Cartier R. Outcome with high blood lactate levels during cardiopulmonary bypass in adult cardiac operation. Ann Thorac Surg. 2000 Dec;70(6):2082-6. doi: 10.1016/s0003-4975(00)02160-3. PMID 11156124
- [Background] Van Erp AC, Rebolledo RA, Hoeksma D, Jespersen NR, Ottens PJ, Norregaard R, Pedersen M, Laustsen C, Burgerhof JGM, Wolters JC, Ciapaite J, Botker HE, Leuvenink HGD, Jespersen B. Organ-specific responses during brain death: increased aerobic metabolism in the liver and anaerobic metabolism with decreased perfusion in the kidneys. Sci Rep. 2018 Mar 13;8(1):4405. doi: 10.1038/s41598-018-22689-9. PMID 29535334
- [Background] Fletcher NM, Awonuga AO, Neubauer BR, Abusamaan MS, Saed MG, Diamond MP, Saed GM. Shifting anaerobic to aerobic metabolism stimulates apoptosis through modulation of redox balance: potential intervention in the pathogenesis of postoperative adhesions. Fertil Steril. 2015 Oct;104(4):1022-1029. doi: 10.1016/j.fertnstert.2015.06.041. Epub 2015 Jul 26. PMID 26215756
- [Background] Ross JM, Oberg J, Brene S, Coppotelli G, Terzioglu M, Pernold K, Goiny M, Sitnikov R, Kehr J, Trifunovic A, Larsson NG, Hoffer BJ, Olson L. High brain lactate is a hallmark of aging and caused by a shift in the lactate dehydrogenase A/B ratio. Proc Natl Acad Sci U S A. 2010 Nov 16;107(46):20087-92. doi: 10.1073/pnas.1008189107. Epub 2010 Nov 1. PMID 21041631
- [Background] Myers J, Ashley E. Dangerous curves. A perspective on exercise, lactate, and the anaerobic threshold. Chest. 1997 Mar;111(3):787-95. doi: 10.1378/chest.111.3.787. PMID 9118720
- [Background] Navarro D, Zwingmann C, Hazell AS, Butterworth RF. Brain lactate synthesis in thiamine deficiency: a re-evaluation using 1H-13C nuclear magnetic resonance spectroscopy. J Neurosci Res. 2005 Jan 1-15;79(1-2):33-41. doi: 10.1002/jnr.20290. PMID 15573405
- [Background] Ba A. Metabolic and structural role of thiamine in nervous tissues. Cell Mol Neurobiol. 2008 Nov;28(7):923-31. doi: 10.1007/s10571-008-9297-7. Epub 2008 Jul 19. PMID 18642074
- [Background] Harrigan GG, Maguire G, Boros L. Metabolomics in alcohol research and drug development. Alcohol Res Health. 2008;31(1):26-35. PMID 23584749
- [Background] Donnino MW, Miller J, Goyal N, Loomba M, Sankey SS, Dolcourt B, Sherwin R, Otero R, Wira C. Effective lactate clearance is associated with improved outcome in post-cardiac arrest patients. Resuscitation. 2007 Nov;75(2):229-34. doi: 10.1016/j.resuscitation.2007.03.021. Epub 2007 Jun 20. PMID 17583412
- [Background] Campbell CH. Lacticacidosis and thiamine deficiency. Lancet. 1984 Dec 1;2(8414):1282. doi: 10.1016/s0140-6736(84)92835-6. No abstract available. PMID 6150313
- [Background] Crook MA. Chapter 6 - Methods for assessment of Thiamine (Vitamin B1). In: Harrington D, ed. Laboratory Assessment of Vitamin Status. Academic Press; 2019:149-64.
- [Background] Thomson AD, Guerrini I, Marshall EJ. Wernicke's encephalopathy: role of thiamine. Pract Gastroenterol 33: 21-30, 2009.
- [Background] Sullivan EV, Fama R. Wernicke's encephalopathy and Korsakoff's syndrome revisited. Neuropsychol Rev. 2012 Jun;22(2):69-71. doi: 10.1007/s11065-012-9205-2. Epub 2012 May 16. No abstract available. PMID 22588370
- [Background] Butterworth RF. Effects of thiamine deficiency on brain metabolism: implications for the pathogenesis of the Wernicke-Korsakoff syndrome. Alcohol Alcohol. 1989;24(4):271-9. doi: 10.1093/oxfordjournals.alcalc.a044913. PMID 2675860
- [Background] Sriram K, Manzanares W, Joseph K. Thiamine in nutrition therapy. Nutr Clin Pract. 2012 Feb;27(1):41-50. doi: 10.1177/0884533611426149. Epub 2012 Jan 4. PMID 22223666
- [Background] Attaluri P, Castillo A, Edriss H, Nugent K. Thiamine Deficiency: An Important Consideration in Critically Ill Patients. Am J Med Sci. 2018 Oct;356(4):382-390. doi: 10.1016/j.amjms.2018.06.015. Epub 2018 Jun 21. PMID 30146080
- [Background] Page GL, Laight D, Cummings MH. Thiamine deficiency in diabetes mellitus and the impact of thiamine replacement on glucose metabolism and vascular disease. Int J Clin Pract. 2011 Jun;65(6):684-90. doi: 10.1111/j.1742-1241.2011.02680.x. PMID 21564442
- [Background] DiNicolantonio JJ, Liu J, O'Keefe JH. Thiamine and Cardiovascular Disease: A Literature Review. Prog Cardiovasc Dis. 2018 May-Jun;61(1):27-32. doi: 10.1016/j.pcad.2018.01.009. Epub 2018 Jan 31. PMID 29360523
- [Background] Levy WC, Soine LA, Huth MM, Fishbein DP. Thiamine deficiency in congestive heart failure. Am J Med. 1992 Dec;93(6):705-6. doi: 10.1016/0002-9343(92)90212-t. No abstract available. PMID 1466372
- [Background] Jain A, Mehta R, Al-Ani M, Hill JA, Winchester DE. Determining the Role of Thiamine Deficiency in Systolic Heart Failure: A Meta-Analysis and Systematic Review. J Card Fail. 2015 Dec;21(12):1000-7. doi: 10.1016/j.cardfail.2015.10.005. Epub 2015 Oct 20. PMID 26497757
- [Background] Lomivorotov VV, Moroz G, Ismoilov S, Shmyrev V, Efremov S, Abubakirov M, Batalov V, Landoni G, Lembo R, Bogachev-Prokophiev A, Sapegin A, Bellomo R. Sustained High-dose Thiamine Supplementation in High-risk Cardiac Patients Undergoing Cardiopulmonary Bypass: A Pilot Feasibility Study (The APPLY trial). J Cardiothorac Vasc Anesth. 2020 Mar;34(3):594-600. doi: 10.1053/j.jvca.2019.08.044. Epub 2019 Sep 4. PMID 31558398
- [Background] Brady JA, Rock CL, Horneffer MR. Thiamin status, diuretic medications, and the management of congestive heart failure. J Am Diet Assoc. 1995 May;95(5):541-4. doi: 10.1016/S0002-8223(95)00148-4. PMID 7722187
- [Background] Pfitzenmeyer P, Guilland JC, d'Athis P, Petit-Marnier C, Gaudet M. Thiamine status of elderly patients with cardiac failure including the effects of supplementation. Int J Vitam Nutr Res. 1994;64(2):113-8. PMID 7960489
- [Background] Zheng Y, Li D, Zeng N, Guo H, Li H, Shen S. Trends of antihypertensive agents in patients with hypertension and coronary artery disease in a tertiary hospital of China. Int J Clin Pharm. 2020 Apr;42(2):482-488. doi: 10.1007/s11096-020-00986-6. Epub 2020 Feb 20. PMID 32078105
- [Background] Li Q, Chen Q, Zhang H, Xu Z, Wang X, Pang J, Ma J, Ling W, Li D. Associations of serum magnesium levels and calcium-magnesium ratios with mortality in patients with coronary artery disease. Diabetes Metab. 2020 Oct;46(5):384-391. doi: 10.1016/j.diabet.2019.12.003. Epub 2019 Dec 20. PMID 31870835
- [Background] Nardin M, Verdoia M, Negro F, Rolla R, Tonon F, De Luca G. Impact of active smoking on the immature platelet fraction and its relationship with the extent of coronary artery disease. Eur J Clin Invest. 2020 Feb;50(2):e13181. doi: 10.1111/eci.13181. Epub 2020 Jan 18. PMID 31659742
- [Background] Inaguma D, Koide S, Takahashi K, Hayashi H, Hasegawa M, Yuzawa Y. Relationship between history of coronary heart disease at dialysis initiation and onset of events associated with heart disease: a propensity-matched analysis of a prospective cohort study. BMC Nephrol. 2017 Feb 28;18(1):79. doi: 10.1186/s12882-017-0495-8. PMID 28245790
- [Background] Tong J, Liu M, Li H, Luo Z, Zhong X, Huang J, Liu R, He F, Fu J. Mortality and Associated Risk Factors in Dialysis Patients with Cardiovascular Disease. Kidney Blood Press Res. 2016;41(4):479-87. doi: 10.1159/000443449. Epub 2016 Jul 20. PMID 27434642
- [Background] Chionh CY, Clementi A, Poh CB, Finkelstein FO, Cruz DN. The use of peritoneal dialysis in heart failure: A systematic review. Perit Dial Int. 2020 Nov;40(6):527-539. doi: 10.1177/0896860819895198. Epub 2020 Jan 13. PMID 32063182
- [Background] Francois K, Ronco C, Bargman JM. Peritoneal Dialysis for Chronic Congestive Heart Failure. Blood Purif. 2015;40(1):45-52. doi: 10.1159/000430084. Epub 2015 Jun 24. PMID 26111872
- [Background] Grossekettler L, Schmack B, Meyer K, Brockmann C, Wanninger R, Kreusser MM, Frankenstein L, Kihm LP, Zeier M, Katus HA, Remppis A, Schwenger V. Peritoneal dialysis as therapeutic option in heart failure patients. ESC Heart Fail. 2019 Apr;6(2):271-279. doi: 10.1002/ehf2.12411. Epub 2019 Feb 27. PMID 30815994
- [Background] Suter PM, Vetter W. Diuretics and vitamin B1: are diuretics a risk factor for thiamin malnutrition? Nutr Rev. 2000 Oct;58(10):319-23. doi: 10.1111/j.1753-4887.2000.tb01827.x. PMID 11127971
- [Background] Hung SC, Hung SH, Tarng DC, Yang WC, Chen TW, Huang TP. Thiamine deficiency and unexplained encephalopathy in hemodialysis and peritoneal dialysis patients. Am J Kidney Dis. 2001 Nov;38(5):941-7. doi: 10.1053/ajkd.2001.28578. PMID 11684545
- [Background] Amrein K, Ribitsch W, Otto R, Worm HC, Stauber RE. Severe lactic acidosis reversed by thiamine within 24 hours. Crit Care. 2011;15(6):457. doi: 10.1186/cc10495. Epub 2011 Dec 1. No abstract available. PMID 22129138
- [Background] Oriot D, Wood C, Gottesman R, Huault G. Severe lactic acidosis related to acute thiamine deficiency. JPEN J Parenter Enteral Nutr. 1991 Jan-Feb;15(1):105-9. doi: 10.1177/0148607191015001105. PMID 1901099
- [Background] Madl C, Kranz A, Liebisch B, Traindl O, Lenz K, Druml W. Lactic acidosis in thiamine deficiency. Clin Nutr. 1993 Apr;12(2):108-11. doi: 10.1016/0261-5614(93)90060-h. PMID 16843296
- [Background] Woolum JA, Abner EL, Kelly A, Thompson Bastin ML, Morris PE, Flannery AH. Effect of Thiamine Administration on Lactate Clearance and Mortality in Patients With Septic Shock. Crit Care Med. 2018 Nov;46(11):1747-1752. doi: 10.1097/CCM.0000000000003311. PMID 30028362
- [Background] Luger M, Hiesmayr M, Koppel P, Sima B, Ranz I, Weiss C, Konig J, Luger E, Kruschitz R, Ludvik B, Schindler K. Influence of intravenous thiamine supplementation on blood lactate concentration prior to cardiac surgery: A double-blinded, randomised controlled pilot study. Eur J Anaesthesiol. 2015 Aug;32(8):543-8. doi: 10.1097/EJA.0000000000000205. PMID 26066773
- [Background] Vacas S, Degos V, Feng X, Maze M. The neuroinflammatory response of postoperative cognitive decline. Br Med Bull. 2013;106(1):161-78. doi: 10.1093/bmb/ldt006. Epub 2013 Apr 4. PMID 23558082
- [Background] Atkinson TM, Konold TR, Glutting JJ. Patterns of memory: a normative taxonomy of the Wide Range Assessment of Memory and Learning-Second Edition (WRAML-2). J Int Neuropsychol Soc. 2008 Sep;14(5):869-77. doi: 10.1017/S1355617708081137. PMID 18764982
- [Background] Pike NA, Poulsen MK, Woo MA. Validity of the Montreal Cognitive Assessment Screener in Adolescents and Young Adults With and Without Congenital Heart Disease. Nurs Res. 2017 May/Jun;66(3):222-230. doi: 10.1097/NNR.0000000000000192. PMID 28448372
- [Background] Gil L, Ruiz de Sanchez C, Gil F, Romero SJ, Pretelt Burgos F. Validation of the Montreal Cognitive Assessment (MoCA) in Spanish as a screening tool for mild cognitive impairment and mild dementia in patients over 65 years old in Bogota, Colombia. Int J Geriatr Psychiatry. 2015 Jun;30(6):655-62. doi: 10.1002/gps.4199. Epub 2014 Oct 16. PMID 25320026
- [Background] Cicione A, Brassetti A, Lombardo R, Franco A, Turchi B, D'Annunzio S, Nacchia A, Tubaro A, Simone G, De Nunzio C. Metabolic Syndrome and Physical Inactivity May Be Shared Etiological Agents of Prostate Cancer and Coronary Heart Diseases. Cancers (Basel). 2022 Feb 14;14(4):936. doi: 10.3390/cancers14040936. PMID 35205684
- [Background] Pike NA, Woo MA, Poulsen MK, Evangelista W, Faire D, Halnon NJ, Lewis AB, Kumar R. Predictors of Memory Deficits in Adolescents and Young Adults with Congenital Heart Disease Compared to Healthy Controls. Front Pediatr. 2016 Oct 31;4:117. doi: 10.3389/fped.2016.00117. eCollection 2016. PMID 27843890
- [Background] Cook CC. Prevention and treatment of Wernicke-Korsakoff syndrome. Alcohol Alcohol Suppl. 2000 May-Jun;35(1):19-20. doi: 10.1093/alcalc/35.supplement_1.19. PMID 11304070
- [Background] Thomson AD, Cook CC. Parenteral thiamine and Wernicke's encephalopathy: the balance of risks and perception of concern. Alcohol Alcohol. 1997 May-Jun;32(3):207-9. doi: 10.1093/oxfordjournals.alcalc.a008259. PMID 9199720
- [Background] Thomson AD, Cook CC, Touquet R, Henry JA; Royal College of Physicians, London. The Royal College of Physicians report on alcohol: guidelines for managing Wernicke's encephalopathy in the accident and Emergency Department. Alcohol Alcohol. 2002 Nov-Dec;37(6):513-21. doi: 10.1093/alcalc/37.6.513. PMID 12414541
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Singh S, Roy B, Halnon NJ, Lewis AB, Woo MA, Pike NA, Kumar R. Regional brain changes in autonomic, mood, and cognitive control areas in adolescents with single ventricle heart disease. International Society for Magnetic Resonance in Medicine Annual Meeting, Paris, France, June 16-21, 2018: 2018.
- [Background] Michalowska I, Furmanek MI, Smaga E, Juraszynski Z, Zielinski T, Chelstowska S, Kusmierczyk M, Szpakowski E, Mierzynska A, Walecki JM. Evaluation of brain lesions in patients after coronary artery bypass grafting using MRI with the emphasis on susceptibility-weighted imaging. Kardiochir Torakochirurgia Pol. 2015 Mar;12(1):1-7. doi: 10.5114/kitp.2015.50560. Epub 2015 Mar 31. PMID 26336470
- [Background] Kumar R, Delshad S, Macey PM, Woo MA, Harper RM. Development of T2-relaxation values in regional brain sites during adolescence. Magn Reson Imaging. 2011 Feb;29(2):185-93. doi: 10.1016/j.mri.2010.08.006. Epub 2010 Oct 8. PMID 20933351
- [Background] Kumar R, Nguyen HD, Macey PM, Woo MA, Harper RM. Regional brain axial and radial diffusivity changes during development. J Neurosci Res. 2012 Feb;90(2):346-55. doi: 10.1002/jnr.22757. Epub 2011 Sep 21. PMID 21938736
- [Background] Kumar R, Delshad S, Woo MA, Macey PM, Harper RM. Age-related regional brain T2-relaxation changes in healthy adults. J Magn Reson Imaging. 2012 Feb;35(2):300-8. doi: 10.1002/jmri.22831. Epub 2011 Oct 10. PMID 21987489
- [Background] Tsai JC, Chen CW, Chu H, Yang HL, Chung MH, Liao YM, Chou KR. Comparing the Sensitivity, Specificity, and Predictive Values of the Montreal Cognitive Assessment and Mini-Mental State Examination When Screening People for Mild Cognitive Impairment and Dementia in Chinese Population. Arch Psychiatr Nurs. 2016 Aug;30(4):486-91. doi: 10.1016/j.apnu.2016.01.015. Epub 2016 Jan 21. PMID 27455923
- [Background] Schulz KF, Grimes DA. Unequal group sizes in randomised trials: guarding against guessing. Lancet. 2002 Mar 16;359(9310):966-70. doi: 10.1016/S0140-6736(02)08029-7. PMID 11918933
- [Background] Donnino MW, Andersen LW, Chase M, Berg KM, Tidswell M, Giberson T, Wolfe R, Moskowitz A, Smithline H, Ngo L, Cocchi MN; Center for Resuscitation Science Research Group. Randomized, Double-Blind, Placebo-Controlled Trial of Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. Crit Care Med. 2016 Feb;44(2):360-7. doi: 10.1097/CCM.0000000000001572. PMID 26771781
- [Background] Nishimoto A, Usery J, Winton JC, Twilla J. High-dose Parenteral Thiamine in Treatment of Wernicke's Encephalopathy: Case Series and Review of the Literature. In Vivo. 2017 Jan 2;31(1):121-124. doi: 10.21873/invivo.11034. PMID 28064230
- [Background] Costantini A, Pala MI. Thiamine and fatigue in inflammatory bowel diseases: an open-label pilot study. J Altern Complement Med. 2013 Aug;19(8):704-8. doi: 10.1089/acm.2011.0840. Epub 2013 Feb 4. PMID 23379830
- [Background] Latt N, Dore G. Thiamine in the treatment of Wernicke encephalopathy in patients with alcohol use disorders. Intern Med J. 2014 Sep;44(9):911-5. doi: 10.1111/imj.12522. PMID 25201422
- [Background] Wrenn KD, Murphy F, Slovis CM. A toxicity study of parenteral thiamine hydrochloride. Ann Emerg Med. 1989 Aug;18(8):867-70. doi: 10.1016/s0196-0644(89)80215-x. PMID 2757284
- [Background] Kumar R, Yadav SK, Palomares JA, Park B, Joshi SH, Ogren JA, Macey PM, Fonarow GC, Harper RM, Woo MA. Reduced regional brain cortical thickness in patients with heart failure. PLoS One. 2015 May 11;10(5):e0126595. doi: 10.1371/journal.pone.0126595. eCollection 2015. PMID 25962164
- [Background] Tummala S, Palomares J, Kang DW, Park B, Woo MA, Harper RM, Kumar R. Global and Regional Brain Non-Gaussian Diffusion Changes in Newly Diagnosed Patients with Obstructive Sleep Apnea. Sleep. 2016 Jan 1;39(1):51-7. doi: 10.5665/sleep.5316. PMID 26285005
- [Background] Joosten A, Rinehart J, Bardaji A, Van der Linden P, Jame V, Van Obbergh L, Alexander B, Cannesson M, Vacas S, Liu N, Slama H, Barvais L. Anesthetic Management Using Multiple Closed-loop Systems and Delayed Neurocognitive Recovery: A Randomized Controlled Trial. Anesthesiology. 2020 Feb;132(2):253-266. doi: 10.1097/ALN.0000000000003014. PMID 31939839